CLINICAL TRIAL: NCT03998657
Title: A Continued Access Study to Evaluate Focal MR-Guided Focused Ultrasound Treatment of Localized Intermediate Risk Prostate Lesions
Brief Title: Continued Access of Focal MR-Guided Focused Ultrasound for Localized Intermediate Risk Prostate Lesions
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCa003CA
Record Dates: First submitted 2019-06-17; First posted 2019-06-26 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Exablate Treated Arm (Experimental): Treatment with Exablate Prostate 2100 Type-3 System
  Interventions: Device: Exablate Prostate Treatment

INTERVENTIONS:
Device: Exablate Prostate Treatment — The Exablate system is a non-invasive thermal ablation device that is being used to ablate tissue. The system combines a focused ultrasound surgery (FUS) delivery system and MRI scanner.
  Other Names: Exablate Prostate; Exablate MRgFUS

SUMMARY:
This extended clinical investigation is a multicenter, prospective, single arm study intended to provide continued access of the Exablate Model 2100 device (Exablate Prostate) to patients for treatment of prostate lesions and collect additional safety and effectiveness data during the 510(k) preparation and review period.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven adenocarcinoma of the prostate
* Intermediate risk, organ-confined prostate cancer (T1a up to T2b) and voluntarily chooses Exablate, who may currently be on watchful waiting or active surveillance and not in need of imminent radical therapy
* Up to 2 MRI visible Gleason 7 confirmed on mapping prostate biopsy that Investigator deems treatable within a single treatment session; may have secondary Gleason 6 on ipsilateral or contralateral side confirmed with biopsy and/or MRI
* PSA less than or equal to 20ng/mL

Exclusion Criteria:

* Evidence of distant prostate cancer including lymph node involvement and/or metastasis of cancer
* Subject undergoing androgen deprivation therapy, initiating any new medication that can affect PSA, or history of bilateral orchiectomy
* Active bladder cancer, active UTI, or untreated prostatitis
* Untreated urethral stricture/bladder neck contracture
* Prostate-specific chemotherapy, brachytherapy, cryotherapy, photodynamic therapy, radical prostatectomy, or focal therapy (excluding FUS); or any prior radiation therapy to the pelvis for prostate cancer or any other malignancy
* Subjects with pathology or implants that may adversely impact treatment due to acoustics, imaging, or safe probe insertion
* Subject not able or willing to tolerate the required prolonged stationary supine position during treatment
* Contraindications to MRI

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Males only
Enrollment: 14 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of device/procedure-related complications following treatment | 12 months
  Safety will be evaluated by incidence and severity of device/procedure-related complications following treatment. Adverse events will be recorded and categorized according to severity and relationship to the biopsy procedure, the Exablate procedure, or to the Exablate device. They will be classified based on body system, severity, and frequency.
Proportions of treated subjects reporting negative Gleason 7 biopsy within the prostate biopsy treatment area. | 6 months
  Effectiveness will be evaluated by targeted lesion control based on biopsy results. Proportions of treated subjects reporting negative Gleason 7 biopsy within the treatment area and/or MRI verification of index lesion(s) ablation. PSA results and validated subject-reported questionnaires will be summarized.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Stanford University School of Medicine, Stanford, California
  - Sperling Prostate Center, Delray Beach, Florida
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Memorial Sloan-Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: No